CLINICAL TRIAL: NCT06762509
Title: The Clinical Study of Botulinum Toxin Type A Injection in the Treatment of Wilson Disease
Acronym: WD
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jun Li, Chief physician, The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Other Study IDs: BTTA; gxgwfx2021028 (Other Grant/Funding Number: Department of education, Anhui Province)
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Wilson Disease
Keywords: botulinum toxin type A; wilson disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- botulinum toxin type A: Enrolled patients were given basic copper discharge treatment, including sodium dimercaptopropyl sulfonate injection, dimercaptosuccinic acid capsules, zinc gluconate tablets, benzoxol hydrochloride tablets, etc. Local injection of botulinum toxin type A was given at the time of enrollment.
  Placebo Comparator: Control group Arm Description: Enrolled patients were treated with DMPS basic copper expulsion therapy, including sodium dithioglycolate injection, dithioglycolic acid capsules, zinc gluconate tablets, benzoxol hydrochloride tablets, etc.
  Interventions: Drug: Botulinum toxin type A
- Enrolled patients were treated with DMPS basic copper expulsion therapy: Enrolled patients were treated with DMPS basic copper expulsion therapy, including sodium dithioglycolate injection, dithioglycolic acid capsules, zinc gluconate tablets, benzoxol hydrochloride tablets, etc.

INTERVENTIONS:
Drug: Botulinum toxin type A — Local injection of botulinum toxin type A was given at the time of enrollment
  Groups: botulinum toxin type A

SUMMARY:
In order to expand the treatment of Wilson disease and improve the quality of life of patients with Wilson's disease, the clinical effect of botulinum toxin type A injection on Wilson's disease was discussed.

ELIGIBILITY:
Inclusion Criteria：1.Conform to the diagnosis of "2012 European Liver Study Guidelines for Diagnosis and Treatment of hepatolenticular degeneration". 2. Aged from 15 to 65 years.

Exclusion Criteria:Non-Wilson's disease

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Unified Dystonia Rating Scale(UDRS) | 4 weeks
  Unified Dystonia Rating Scale(UDRS),Higher scores mean a worse outcome.
Unified Wilson's Disease Rating Scale(UWDRS) | 4 weeks
  Unified Wilson's Disease Rating Scale(UWDRS).Higher scores mean a worse outcome
Numeric Rating Scales(NRS) | 4 weeks
  Numeric Rating Scales(NRS),Higher scores mean a worse outcome
Activity of Daily Living Scale(ADL) | 4 weeks
  Activity of Daily Living Scale,Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, #117 Meishan Street, Shushan District Hefei 230037, China, Hefei, China

IPD SHARING:
Plan to Share IPD: Undecided